CLINICAL TRIAL: NCT05167864
Title: A Randomized Prospective Evaluation of Four Injectable Neuromodulators in the Glabella Area
Brief Title: Evaluation of Four Injectable Neuromodulators in the Glabella Area Glabella Area
Acronym: JBDX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 849045
Record Dates: First submitted 2021-12-03; First posted 2021-12-22 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Cosmetic Techniques
Keywords: minimally invasive procedures; neurotoxins; cosmetic; Botox; eyebrow area; glabella; Dysport; Jeuveau; Xeomin; forehead; cosmetic injections; facial rejuvenation; wrinkle reduction
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections; abobotulinumtoxinA; incobotulinumtoxinA; prabotulinumtoxin A

STUDY DESIGN:
Intervention Model Description: randomized controlled trial in which patients will be randomly assigned into one of four groups
Who Masked: Participant, Care Provider
Masking Description: blinding of participant and provider administering the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- OnabotulinumtoxinA (Active Comparator): Botox
  Interventions: Drug: Onabotulinumtoxina for Injection
- AbobotulinumtoxinA (Active Comparator): Dysport
  Interventions: Drug: Abobotulinumtoxina for Injection
- IncobotulinumtoxinA (Active Comparator): Xeomin
  Interventions: Drug: IncobotulinumtoxinA for Injection
- PrabotulinumtoxinA (Active Comparator): Jeuveau
  Interventions: Drug: PrabotulinumtoxinA for Injection

INTERVENTIONS:
Drug: Onabotulinumtoxina for Injection — cosmetic injection into the glabella area (eyebrow area)
  Other Names: Botox
  Arms: OnabotulinumtoxinA
Drug: Abobotulinumtoxina for Injection — cosmetic injection into the glabella area (eyebrow area)
  Other Names: Dysport
  Arms: AbobotulinumtoxinA
Drug: IncobotulinumtoxinA for Injection — cosmetic injection into the glabella area (eyebrow area)
  Other Names: Xeomin
  Arms: IncobotulinumtoxinA
Drug: PrabotulinumtoxinA for Injection — cosmetic injection into the glabella area (eyebrow area)
  Other Names: Jeuveau
  Arms: PrabotulinumtoxinA

SUMMARY:
The purpose of the study is to use 3D imaging to evaluate the effects of four FDA approved neuromodulators on facial lines, wrinkles and animation. Participation is available to women who have never had a cosmetic procedure above the malar region nor a treatment with a neuromodulator within 12 months. All subjects will undergo 3D imaging using the VECTRA M3 (Canfield Scientific, Inc, Fairfield, NJ) prior to treatment with a neuromodulator in order to determine their baseline dimensions. Imaging will be repeated post injection to determine change over time.

DETAILED DESCRIPTION:
This study is a randomized controlled trial in which patients will be randomly assigned into one of four groups: those receiving onabotulinumtoxinA (Botox, Allergan, Irvine, California), abobotulinumtoxinA (Dysport, Ispen Biopharmacueticals Inc.Cambridge, MA), incobotulinumtoxinA (Xeomin, Raleigh, NC) or prabotulinumtoxinA (Jeuveau, Evolus, Newport Beach, California). Each patient will receive FDA approved dosages in which they are assigned in to treat rhytids within the glabella, as per FDA approved indications. All injections will be performed by a blinded single trained physician according to a preset injection plan per FDA approved administration guidelines. Prior to injection patients will be imaged with 3-dimensional photogrammetry. All pre-procedure images will be evaluated for absolute strain performing two types of facial animation: 1) relaxed, and 2) frowning. Subjects will return Day 3, 30, 90, and 180, post intervention for re-imaging with the same expressions. Strain will be calculated using the same metrics.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 30-65 years of age
* Interested in glabellar injections to reduce rhytids and facial strain
* Participants must sign the informed consent form

Exclusion Criteria:

* Females under 30 or above 65 years of age
* Males
* Those who have received glabellar injections for rhytids <12 months
* Underwent cosmetic surgical procedure above the malar region
* Those with a condition that affects facial expression, such as prior stroke

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Lemdani MS, Honig SE, Habarth-Morales TE, Davis HD, Niu EF, Ewing JN, Broach RB, Serletti JM, Percec I. Comparison of Botulinum Toxin A Formulations for Glabellar Strain Treatment in Women: A Double-Blind Randomized Clinical Trial. JAMA Dermatol. 2025 Jul 1;161(7):723-730. doi: 10.1001/jamadermatol.2025.1335. PMID 40434770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OnabotulinumtoxinA | AbobotulinumtoxinA | IncobotulinumtoxinA | PrabotulinumtoxinA
Started | 35 | 36 | 36 | 36
Completed | 28 | 30 | 29 | 27
Not Completed | 7 | 6 | 7 | 9
Not completed — Lost to Follow-up | 7 | 6 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA | AbobotulinumtoxinA | IncobotulinumtoxinA | PrabotulinumtoxinA | Total
Number analyzed (Participants) | 35 | 36 | 36 | 36 | 143
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (10.3) | 44.2 (9.5) | 42.5 (10.6) | 41.9 (8.9) | 43.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 36 | 36 | 143
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 2 | 3 | 2 | 0 | 7
  White/Caucasian | 29 | 30 | 33 | 33 | 125
  Asian | 1 | 3 | 0 | 2 | 6
  Declined to Answer | 3 | 0 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: the Change in Dynamic Strain in the Glabella Area After Injection Over Time
Description: The change in dynamic strain of the glabella area after injection using 3D facial imaging measurements over time At each visit two images were captured, one neutral and one dynamic. The neutral face was relaxed and served as a reference while the dynamic face was the subject's expression when asked to furrow their glabella by frowning (compressed face). A decrease in strain indicates reduced compression, as there is a smaller difference between the neutral face and the dynamic, or compressed, face.
Time Frame: day 3, day 30, day 90, day 180
Population: the change in dynamic strain is determined by measurements changes from two 3D images, if the images were not captured or the images were deemed unanalyzable then the population analyzed varies from the participant count.
Measure: Mean (Standard Deviation); unit: percent difference of neutral+dyanamic
Arm/Group | OnabotulinumtoxinA | AbobotulinumtoxinA | IncobotulinumtoxinA | PrabotulinumtoxinA
Number analyzed (Participants) | 34 | 34 | 34 | 36
percent difference of neutral+dyanamic
  Day 3 | 6.4 (5.0) | 10.9 (5.2) | 6.6 (5.6) | 8.9 (4.6)
  Day 30 | 8.6 (5.4) | 10.6 (6.2) | 9.2 (5.7) | 10.4 (4.3)
  Day 90 | 4.5 (4.6) | 5.7 (5.2) | 3.6 (5.3) | 5.2 (3.7)
  Day 180 | 0.18 (4.1) | 2.3 (5.6) | 2.6 (4.7) | 3.1 (4.4)

2. Secondary Outcome: Correlation Patient Reported Satisfaction (FACE-Q) to the Degree of Dynamic Strain Overtime
Description: Correlation of patient reported satisfaction (FACE-Q) to the degree of dynamic strain overtime. Correlation is determined at each time point post intervention Day 3, Day 30, Day 90 and Day 180.
Time Frame: baseline, day 3, day 30, day 90, day 180
Population: population of who answered the FACE-Q can be analyzed
Measure: Mean (Standard Error); unit: correlation coefficient
Arm/Group | OnabotulinumtoxinA | AbobotulinumtoxinA | IncobotulinumtoxinA | PrabotulinumtoxinA
Number analyzed (Participants) | 34 | 34 | 34 | 36
correlation coefficient
  Appraisal of Lines: Forehead Day 3 | -0.0870 (0.057) | -0.013 (0.052) | 0.049 (0.661) | -0.095 (0.045)
  Appraisal of Lines: Forehead Day 30 | 0.033 (0.492) | -0.018 (0.061) | -0.338 (0.055) | -0.0877 (0.046)
  Appraisal of Lines: Forehead Day 90 | 0.0327 (0.053) | -0.012 (0.039) | 0.021 (0.053) | -0.039 (.045)
  Appraisal of Lines: Forehead Day 180 | -0.086 (0.048) | -0.065 (0.064) | -0.071 (0.0501) | -0.014 (0.090)
  Satisfaction with Forehead Day 3 | -0.059 (0.086) | -0.010 (0083) | 0.033 (0.083) | -0.059 (0.051)
  Satisfaction with Forehead Day 30 | 0.015 (0.066) | 0.075 (0.066) | -0.002 (0.070) | -0.028 (0.041)
  Satisfaction with Forehead Day 90 | -0.028 (0.087) | -0.042 (0.53) | 0.015 (0.069) | 0.015 (0.069)
  Satisfaction with Forehead Day 180 | -0.053 (0.081) | -0.010 (0.044) | -0.031 (0.066) | 0.111 (0.063)
  Appraisal of Lines between Eyebrows Day 3 | -0.015 (0.031) | 0.046 (0.047) | 0.064 (0.043) | -0.038 (0.041)
  Appraisal of Lines between Eyebrows Day 30 | 0.025 (0.315) | 0.009 (0.045) | 0.048 (0.047) | 0.027 (0.026)
  Appraisal of Lines between Eyebrows Day 90 | 0.008 (0.053) | 0.030 (0.040) | -0.015 (0.046) | 0.009 (0.028)
  Appraisal of Lines between Eyebrows Day 180 | 0.024 (0.041) | 0.015 (0.069) | -0.133 (0.041) | 0.034 (0.043)
Statistical Analysis 1: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.13519, Wilcoxon signed-rank sum test; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement of line in the forehead post injection day 3
Statistical Analysis 2: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.8556, Wilcoxon signed-rank sum test; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.46943, Wilcoxon signed-rank test; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.0449, Wilcoxon signed-rank sum test; [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.504, Wilcoxon signed-rank sum test; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement of line in the forehead post injection day 30
Statistical Analysis 6: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.772193, Wilcoxon signed-rank sum test; [other analysis details as in outcome 2, analysis 5]
Statistical Analysis 7: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.5414, Wilcoxon signed-rank sum test; [other analysis details as in outcome 2, analysis 5]
Statistical Analysis 8: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.070, Wilcoxon signed-rank sum test; [other analysis details as in outcome 2, analysis 5]
Statistical Analysis 9: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.546, Wilcoxon signed rank sum test; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement of line in the forehead post injection day 90
Statistical Analysis 10: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.756, Wilcoxon signed rank sum test; [other analysis details as in outcome 2, analysis 9]
Statistical Analysis 11: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.700, Wilcoxon signed rank sum test; [other analysis details as in outcome 2, analysis 9]
Statistical Analysis 12: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.397, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 9]
Statistical Analysis 13: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.093, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement of line in the forehead post injection day 180
Statistical Analysis 14: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.323, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 13]
Statistical Analysis 15: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.182, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) tothe patient satisfaction improvement of line in the forehead post injection day 180
Statistical Analysis 16: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.880, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 13]
Statistical Analysis 17: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.496, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) tothe patient satisfaction improvement in the forehead post injection day 3
Statistical Analysis 18: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.905, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the forehead post injection day 3
Statistical Analysis 19: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.692, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 18]
Statistical Analysis 20: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.262, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 18]
Statistical Analysis 21: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.828, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the forehead post injection day 30
Statistical Analysis 22: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.268, Wilcoxon signed rank sum test; [other analysis details as in outcome 2, analysis 21]
Statistical Analysis 23: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.975, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 21]
Statistical Analysis 24: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.499, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 21]
Statistical Analysis 25: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.750, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the forehead post injection day 90
Statistical Analysis 26: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.433, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 25]
Statistical Analysis 27: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.834, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 25]
Statistical Analysis 28: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.834, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 25]
Statistical Analysis 29: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.526, Wilcoxon signed rank sum test; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the forehead post injection day 180
Statistical Analysis 30: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.816, Wilcoxon singed rank sum; [other analysis details as in outcome 2, analysis 29]
Statistical Analysis 31: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.650, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 29]
Statistical Analysis 32: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.095, wilcoxon rank sum test; [other analysis details as in outcome 2, analysis 29]
Statistical Analysis 33: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.618, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the lines between the eyebrows post injection day 3
Statistical Analysis 34: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.340, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 33]
Statistical Analysis 35: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.150, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 33]
Statistical Analysis 36: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.361, Wilcoxon signed rank sum test; [other analysis details as in outcome 2, analysis 33]
Statistical Analysis 37: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.428, wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the lines between the eyebrows post injection day 30
Statistical Analysis 38: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.834, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 37]
Statistical Analysis 39: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.318, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 37]
Statistical Analysis 40: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.311, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 37]
Statistical Analysis 41: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.885, Wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the lines between the eyebrows post injection day 90
Statistical Analysis 42: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.457, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 41]
Statistical Analysis 43: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.745, Wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 41]
Statistical Analysis 44: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.757, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 41]
Statistical Analysis 45: Comparison: OnabotulinumtoxinA; Test type: Superiority; p = 0.562, wilcoxon signed rank sum; the correlation of dynamic strain (decreased compression) to the patient satisfaction improvement in the lines between the eyebrows post injection day 180
Statistical Analysis 46: Comparison: AbobotulinumtoxinA; Test type: Superiority; p = 0.828, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 45]
Statistical Analysis 47: Comparison: IncobotulinumtoxinA; Test type: Superiority; p = 0.005, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 45]
Statistical Analysis 48: Comparison: PrabotulinumtoxinA; Test type: Superiority; p = 0.437, wilcoxon signed rank sum; [other analysis details as in outcome 2, analysis 45]

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | OnabotulinumtoxinA | AbobotulinumtoxinA | IncobotulinumtoxinA | PrabotulinumtoxinA
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/36 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT05167864/Prot_SAP_000.pdf